CLINICAL TRIAL: NCT00768144
Title: A Phase II Trial of Sunitinib in Recurrent and Refractory Ovarian, Fallopian Tube and Peritoneal Carcinoma
Brief Title: Sunitinib in Recurrent and Refractory Ovarian, Fallopian Tube and Peritoneal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana M. Campos, MD, Medical Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-056
Record Dates: First submitted 2008-09-29; First posted 2008-10-07 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Sutent; sunitinib
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): Patients received oral Sunitinib at the daily dose of 37.5 mg continuously over a 28- day treatment cycle. Treatment continued until clinical or radiological evidence of progressive disease or excessive toxicity.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib
  Other Names: Sutent

SUMMARY:
The purpose of this study is to determine the effectiveness of sunitinib on participants with ovarian, fallopian tube or peritoneal cancer. Sunitinib is a newly discovered drug that may stop cancer cells from growing by blocking the blood supply to the tumor.

DETAILED DESCRIPTION:
This study used a two-stage design to evaluate efficacy of sunitinib based on overall response (OR) defined as complete response (CR) or partial response (PR). The null and alternative OR rate were 5% and 20%. If one or more patients enrolled in the stage one cohort (n=17 patients) achieved PR or better than accrual would proceed to stage two (n=18 patients). There was 42% probability of stopping the trial at stage one if the true OR rate was 5%. With 35 patients, this design had 85% power to detect the 15% difference in OR rates assuming 2-sided type I error rate of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed epithelial ovarian, fallopian tube or peritoneal cancer
* Recurrent or refractory disease
* Measurable disease, defined by RECIST
* 0 to 3 prior cytotoxic chemotherapy or biologic regimens for metastatic disease
* Adverse events related to prior tumor-specific therapy must have resolved to less than or equal to grade 1 prior to study entry
* Ability to swallow oral medications
* 18 years of age or older
* ECOG Performance status must be 0-2
* Normal organ and marrow function as outlined in the protocol

Exclusion Criteria:

* Receiving systemic therapy less than 14 days prior to starting sunitinib
* Receiving any other investigational agent
* Received prior sunitinib
* Untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on screening CT or MRI scans
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Evidence of a bleeding diathesis. Major surgery or NCI CTCA 3.0 grade 3 or worse hemorrhage within 4 weeks of starting study treatment
* Ongoing cardiac dysrhythmias of NCI CTCAE version 3.0 grade > 2
* Pre-existing thyroid abnormality, with thyroid function tests that cannot be maintained in the normal range with medication
* Prolonged QTc interval on baseline EKG
* Uncontrolled hypertension
* Patients who are taking cytochrome P450 enzyme-inducing antiepileptic drugs, rifampin, theophylline, ketoconazole, or St. John's wort.
* Psychiatric illness or social situations that wold limit compliance with study requirements
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration
* Pregnant women
* Clinical or radiographical evidence of a small bowel obstruction
* Poor oral intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susana M. Campos, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the GYN Oncology clinics at the DFCI, MGH and BIDMC. Thirty six consenting participants were enrolled over a 19 month period.
Period: Overall Study
Arm/Group | Sunitinib
Started | 36
Completed | 0
Not Completed | 36
Not completed — Adverse Event | 13
Not completed — Progressive Disease | 21
Not completed — Patient or MD Decision to End Treatment | 1
Not completed — Pt Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
Histology [Number; unit: participants]
  Papillary serous | 23
  Endometrioid | 2
  Clear cell | 5
  Mixed Mullerian tumor | 3
  Other (adenocarcinoma/mixed histology) | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Best response on treatment was based on RECIST 1.0 criteria with overall response defined as achieving partial response (PR) or complete response (CR). Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Clinical assessments were performed weekly for first 4 weeks and every 2 wks in subsequent cycles. Disease was evaluated radiologically at baseline, before each odd cycle and at end of trt.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
proportion of participants | .083 [.024 to .210]

2. Secondary Outcome: 16-Week Progression-Free Survival
Description: 16-week progression-free survival is the probability of patients remaining alive and progression-free at 16-weeks from study entry estimated using Kaplan-Meier methods. Patients alive and progression-free at last follow-up are censored. Progressive disease (PD) based on RECIST 1.0 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or equivocal progression of non-target lesions.
Time Frame: Clinical assessments were performed weekly for first 4 weeks and every 2 weeks in subsequent cycles. Disease was evaluated radiologically at baseline, before each odd cycle and at end of treatment.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
probability | .36 [.20 to .52]

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival estimated using Kaplan-Meier methods is defined as the time from registration to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.0 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
weeks | 9.9 [7.1 to 16.4]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment.
Groups:
- Sunitinib: Sunitinib : Taken orally once a day in the evening
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 7/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=36)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — Subject JP: hyperkalemia, grade 4, unrelated to study treatment.
Small bowel obstruction (Gastrointestinal disorders) | 2 (2) — Subject SD: small bowel obstruction, unrelated to study treatment. Subject DM: small bowel obstruction, unrelated to study treatment.
Cerebrovascular accident (Nervous system disorders) | 1 (1) — Subject KG: CVA, possibly related to study treatment.
Allergic reaction (Immune system disorders) | 1 (1) — Subject JH: allergic reaction, grade 3, probably related to study treatment.
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Subject BZG: abdominal pain, possibly related to study treatment.
Death due to progressive disease (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=36)
Hypertension (Vascular disorders) | 36
Fatigue (General disorders) | 36
Vomiting (Gastrointestinal disorders) | 36
Anemia (Blood and lymphatic system disorders) | 8
White blood cell increased (Investigations) | 11
Platelet count decreased (Investigations) | 16
Weight loss (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Diarrhea (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 36
Taste disturbance (Gastrointestinal disorders) | 11
Alkaline phosphatase increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 12
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Proteinuria (Renal and urinary disorders) | 36
Abdominal bloating (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Headache (Nervous system disorders) | 36
Aspartate aminotransferase increased (Investigations) | 12
Creatinine increased (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Mucositis (Gastrointestinal disorders) | 22
Bilirubin increased (Investigations) | 2
Hyponatremia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Depression (Psychiatric disorders) | 2
Alanine aminotransferase increased (Investigations) | 8
Urinary frequency (Renal and urinary disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 6
CNS cerebrovascular ischemia (Vascular disorders) | 2
White blood cell decreased (Investigations) | 4
Neuropathy (Nervous system disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 3
Urine color (Renal and urinary disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Hypothyroidism (Endocrine disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No